CLINICAL TRIAL: NCT03522987
Title: Anxiety and Depression in Epilepsy: A Pilot Epileptologist-Driven Treatment Study
Brief Title: Anxiety and Depression in Epilepsy: A Pilot Treatment Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Decided not to perform the pilot phase
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00048584-1st; 5UL1TR001420-03 (NIH)
Record Dates: First submitted 2018-04-20; First posted 2018-05-14 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2018-07

CONDITIONS: Anxiety; Depression; Epilepsy
Keywords: Neurologic Disorders; Chronic Care; Management; Treatment; SSRI Medication; SNRI Medication; Learning Healthcare System
MeSH Terms: conditions — Anxiety Disorders; Depression; Epilepsy; Nervous System Diseases | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: Epileptologist-driven medication treatment intervention for anxiety and depression, carried out directly in the epilepsy clinic during a regularly scheduled visit and supported by advanced practice provider (APP).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epileptologist-Driven Treatment (Experimental): The intervention will consist of initiating a chronic care management plan in the epilepsy clinic and an initial prescription from the epileptologist for escitalopram 10mg daily. Escitalopram dose adjustment will be made based on biweekly repeated screening of anxiety and depression symptoms, as well as side effects identified on biweekly telephone calls or the 6-week advanced practice provider (APP) follow up visit. Escitalopram dose may be titrated up to a maximum of 20mg daily in 5-10mg increments every 2 weeks for treatment effect, or titrated down to 5mg if needed for adverse effects. If a participant is unable to tolerate escitalopram, then venlafaxine XR 37.5mg will be substituted, to be titrated in a similar manner biweekly based on side effects and anxiety and depression symptoms (with 37.5-75mg increment dose changes and maximum dose of 225mg daily).
  Interventions: Drug: Escitalopram 10mg

INTERVENTIONS:
Drug: Escitalopram 10mg — Participants will be given escitalopram 10mg by mouth daily and will be followed up at 2, 4, 6, 8, and 10 weeks. Medication will be adjusted if side effects occur. If unable to tolerate escitalopram, then venlafaxine XR (Effexor XR) 37.5mg will be substituted.
  Other Names: Lexapro

SUMMARY:
As a potential solution to address high rates of depression and anxiety seen in epilepsy patients and poor mental health care access, this trial aims to carry out treatment for depression and anxiety directly in the epilepsy clinic. Patients that meet eligibility criteria, including significant symptoms of depression and/or anxiety, will be enrolled in the intervention. The intervention will consist of an initial prescription for an FDA-approved medication to treat depression/anxiety and telephone-based chronic care management plan for repeated symptom measurement and side effect surveillance. The purpose of this pre-piloting limited study is to streamline recruitment, intervention and outcome assessment process in preparation for a randomized, controlled pilot of the intervention.

DETAILED DESCRIPTION:
This trial is an innovative learning healthcare system approach to translate the concept of measurement-based depression care into a specialty clinic setting and extend the concept to treat depression and/or anxiety. The neurologist/APP-administered medication intervention utilizes FDA-approved drugs with advantageous features for use in epilepsy (escitalopram and venlafaxine) and a telephone-based chronic care management plan for repeated symptom measurement and side effect surveillance. The proposed intervention may overcome barriers to implementing mental health treatment interventions in generalized clinical settings by using healthcare providers commonly present in specialty clinics (physicians and APPs) along with a billable, best practices chronic care management intervention package. To test this idea, the study team seeks to pilot a feasibility trial of an epileptologist-driven medication treatment intervention for anxiety and depression, carried out directly in the epilepsy clinic during a regularly scheduled visit and supported by advanced practice provider (APP), using epilepsy as a paradigm for chronic medical illness with high prevalence of psychiatric comorbidity. In this limited, intervention only pre-piloting trial, the team will streamline recruitment, intervention, and outcome assessment procedures to prepare for a randomized, controlled pilot of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age 18 or older
* Ability to take oral medication and the willing to adhere to the intervention regimen
* Minimum of 1 prior clinic visit at the Comprehensive Epilepsy Center
* Adequate cognition (MoCA score of 20 or greater)
* Diagnosis of epilepsy: EEG with documented seizure or epileptiform discharges OR non-epileptiform EEG and seizure remission with antiseizure drug OR treating epileptologist's leading clinical impression is epilepsy
* NDDI-E score greater than 15 and/or GAD-7 score greater than or equal to 10

Exclusion Criteria:

* Pregnancy or lactation
* Known allergic reactions to escitalopram or venlafaxine
* Comorbid psychogenic nonepileptic seizures
* Prior psychiatric hospitalization
* Prior suicide attempt
* History of manic or psychotic symptoms (past manic episode (SCID-I), or psychotic symptom screen positive)
* Current treatment by a psychiatrist or counselor/theraptist
* Active suicidality at the time of screening
* Current treatment with buspirone or an SSRI/SNRI/atypical antidepressant (specifically bupropion, fluoxetine, levomilnacipran, citalopram, milnacipran, desvenlafaxine, mirtazapine, duloxetine, paroxetine, escitalopram, sertraline, fluvoxamine, venlafaxine, vilazodone, vortioxetine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Adherence to Intervention | 12 weeks
  Percentage of participants who report taking the prescribed medication at 12 weeks and who have completed at least 2 of the chronic care management scheduled visits (telephone or clinic visit)

SECONDARY OUTCOMES:
Accrual | 12 weeks
  Percentage of patients screened for the trial who are eligible

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Munger Clary, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No